CLINICAL TRIAL: NCT06706687
Title: A Study of the Behavioral Variant of Frontotemporal Dementia and Bipolar Disorder: a Neuroimaging and Epigenetics Integrated Approach
Acronym: DISBAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DISBAND
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Bipolar Disorder; Frontotemporal Dementia, Behavioral Variant
Keywords: Bipolar Disorder (BD); Frontotemporal Dementia, Behavioral Variant (bvFTD); Epigenetics; Neuroimaging; miRNA; Nuclear Magnetic Resonance Imaging (NMR); Nuclear Magnetic Resonance Spectroscopy (1H-MRS); Positron Emission Tomography (PET); Healthy controls (HC)
MeSH Terms: conditions — Bipolar Disorder; Pick Disease of the Brain; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Frontotemporal Dementia, Behavioral Variant (bvFTD) (Other)
  Interventions: Diagnostic Test: DISBAND protocol
- Bipolar Disorder (BD) (Other)
  Interventions: Diagnostic Test: DISBAND protocol
- Healthy controls (HC) (Other)
  Interventions: Diagnostic Test: DISBAND protocol

INTERVENTIONS:
Diagnostic Test: DISBAND protocol — For each participant blood samples will be collected, processed and studied to analyse microRNA expression, more specifically investigating non-coding RNA (ncRNA). Each participant will undergo a multimodal neuroimaging session, composed of structural MRI, 1H-MRS and PET.

SUMMARY:
The aim of this study is to investigate the selective epigenetic modifications and their effect on brain's morphology and functionality in the frontotemporal dementia behavioral variant and bipolar disorder. The open-label, multicentric, interventional case-control study involves the analysis of 3 separate cohorts of patients, partly selected over the course of the past 10 years. More specifically, 80 behavioral variant Frontotemporal Dementia (bvFTD) patients (40, of whom 20 carry G4C2 expansion in the C9orf72 gene, are already available, while 40 will be prospectively recruited), 80 Bipolar Disorder (BD) patients (40, including 20 with early onset and 20 with late onset, are already available, while 40 will be prospectively recruited) and 50 healthy control (HC) subjects (20 of whom are already available from other previously approved studies), will be enrolled in this study.

For each participant a blood sample will be collected, processed, and studied in order analyze the expression of miRNA. Every participant will also undergo Nuclear Magnetic Resonance Imaging (NMR), Nuclear Magnetic Resonance Spectroscopy (1H-MRS), and Positron Emission Tomography (PET) and, lastly, a battery of behavioral scales to explore different cognitive domains will be administered to all participants by a team of psychologists and physicians. The overall estimated duration of the study is 36 months.

DETAILED DESCRIPTION:
Following the inclusion and exclusion criteria, the participants will be recruited and subdivided into three groups:

* bvFTD patients, followed prospectively for at least 2 years. These include bvFTD carriers of G4C2 expansion in the C9orf72 gene (best model of the two diseases because such expansion is widely associated with the development of psychosis)
* BD patients who are part of a cohort of multi affected families (MAF) followed since January 2017 at the Psychiatry Operating Unit of the Policlinico di Milano and who have positive family history of neurodegenerative diseases.
* Healthy subjects who underwent neurocognitive tests at baseline that excluded the presence of dementia and psychiatric diseases.

The investigators will be collecting participants blood samples, which will be processed and analyzed. More specifically, total exosomes will be isolated from 500 microliters of plasma by ExoQuick precipitation solution (SBI). Isolation and purification of NDEs will be performed by ExoFlow purification kit using biotinylated anti-human CD171 (L1CAM) antibody (clone 5G3, Ebiosciences). Total RNA contained in NDEs will be extracted by Total Exosome RNA and Protein Isolation Kit and miRNA expression analysis by TaqMan OpenArray Human Advanced MicroRNA Panel (Thermo Fisher Scientific). Expression analysis of lncRNAs will be conducted by LincFinder Array and inflammatory and autoimmunity arrays (Qiagen).

The participants will also undergo a neuroimaging session, where structural MRI and 1H-MRS sessions will be performed using a 3T MRI scanner available at the Neuroradiology Unit. The 1H-MRS will provide sensitive and reliable assessment of neurochemical changes in specific brain areas. The acquisition voxels will be palced in the dorso- and ventrolateral prefrontal cortex (DLPFC/VLPFC), amygdala, and hippocampus. Finally, an FDG-PET scan will be performed with a Biograph Truepoint 64 PET/TC scanner. T1-weighted and FDG-PET images will be used to explore brain morphological/metabolic differences between the groups. Gray matter and white matter volumes will be estimated locally and compared between groups using voxel-based morphometry. A parallel region of interest comparison (ROIs) will be performed to estimate regional volumes using the Automated Anatomical Labelling (AAL) atlas as a reference, again focusing on the DLPFC/VLPFC, amygdala and hippocampus. Finally, an additional regional analysis based on Freesurfer software will allow the investigators to estimate the cortical thickness, cortical surface area, and cortical gyrification of the Desikan-Killiany atlas regions. All MRI and PET analyses will be performed in the context of a general linear model using a specific software implementation in MATLAB called Statistical Parametric Mapping (SPM).

Lastly, neuroimaging data and ncRNA expression profiles will be used as predictors in the ML analysis. Given the small sample size, initially linear models (e.g., Support Vector Machine) will be used. Later, to improve the predictive power of our models, the investigators will apply the ML method called random forest, a more versatile and powerful classification algorithm, and the XGBoost (eXtreme Gradient Boosting) algorithm. To avoid overfitting of the learning process, a "grid" search of model hyperparameters will be performed. A 5-fold cross-validation will be used to validate the results, with a split between training-tests of 80%-20%.

ELIGIBILITY:
Inclusion Criteria:

* byFTD group: patients of either sex; 18 years of age or older; diagnosis of behavioral variant Frontotemporal Dementia according to current diagnostic criteria; presence of a signed informed consent.
* BD group: patients of either sex; 18 years of age or older; diagnosis of bipolar disorder according to DSM-V criteria; presence of a signed informed consent.
* HC group: patients of either sex; 18 years of age or older; subjects who have gone through the same diagnostic process as patients under suspicion of a central nervous system and/or psychiatric disorder, resulting in the absence of cognitive deficits and mood disorders; presence of a signed informed consent.

Exclusion Criteria:

* Diagnosis of Alzheimer's disease
* Comorbidities interfering with the studied condition (e.g. other neurological diseases or history of substance or alcohol abuse)
* Diseases with an inflammatory component (e.g. autoimmune diseases, tumors)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Identification of ncRNA transcripts and a specific noncoding RNA profile in neuron-derived exosomes | 36 months
  Identification of ncRNA transcripts and a specific noncoding RNA profile in neuron-derived exosomes in patients with bvFTD and BD
Differences in brain structure in terms of white matter volumes | 36 months
  Evaluation of the differences in brain structure in terms of white matter volumes comparing the three groups, using structural MRI
Differences in brain structure in terms of gray matter volumes | 36 months
  Evaluation of the differences in brain structure in terms of gray matter volumes comparing the three groups, using structural MRI
Differences in brain structure in terms of cortical gyrification | 36 months
  Evaluation of the differences in brain structure in terms of cortical gyrification comparing the three groups, using structural MRI
Differences in brain structure in terms of superficial cortical area | 36 months
  Evaluation of the differences in brain structure in terms of superficial cortical area comparing the three groups, using structural MRI
Differences in brain structure in terms of cortical thickness | 36 months
  Evaluation of the differences in brain structure in terms of cortical thickness comparing the three groups, using structural MRI
Differences in brain metabolism | 36 months
  Evaluation of the differences in brain metabolism comparing the three groups, using FDG/PET
Differences in glutamatergic neurotransmission in the prefrontal-limbic cortex | 36 months
  Evaluation of the differences in the glutamatergic neurotransmission of the prefrontal-limbic cortex, comparing the three groups, using 1H-MRS

SECONDARY OUTCOMES:
Creation of a machine learning model | 36 months
  Creation of a machine learning model that could integrate neuroimaging data and miRNA expression data to validate the best candidates identified combining imaging and epigenetic data

CONTACTS AND LOCATIONS:
Overall Officials: Elio Scarpini, Professor, Principal Investigator — UOSD Malattie Neurodegenerative
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galimberti D, Fenoglio C, Serpente M, Villa C, Bonsi R, Arighi A, Fumagalli GG, Del Bo R, Bruni AC, Anfossi M, Clodomiro A, Cupidi C, Nacmias B, Sorbi S, Piaceri I, Bagnoli S, Bessi V, Marcone A, Cerami C, Cappa SF, Filippi M, Agosta F, Magnani G, Comi G, Franceschi M, Rainero I, Giordana MT, Rubino E, Ferrero P, Rogaeva E, Xi Z, Confaloni A, Piscopo P, Bruno G, Talarico G, Cagnin A, Clerici F, Dell'Osso B, Comi GP, Altamura AC, Mariani C, Scarpini E. Autosomal dominant frontotemporal lobar degeneration due to the C9ORF72 hexanucleotide repeat expansion: late-onset psychotic clinical presentation. Biol Psychiatry. 2013 Sep 1;74(5):384-91. doi: 10.1016/j.biopsych.2013.01.031. Epub 2013 Mar 7. PMID 23473366
- [Background] Vieta E, Popovic D, Rosa AR, Sole B, Grande I, Frey BN, Martinez-Aran A, Sanchez-Moreno J, Balanza-Martinez V, Tabares-Seisdedos R, Kapczinski F. The clinical implications of cognitive impairment and allostatic load in bipolar disorder. Eur Psychiatry. 2013 Jan;28(1):21-9. doi: 10.1016/j.eurpsy.2011.11.007. Epub 2012 Apr 24. PMID 22534552
- [Background] Baez S. et al., Neuropsychologia. 2017 Feb 17; S0028-3932(17)30058-1. doi: 10.1016/j.neuropsychologia.2017.02.012.
- [Background] Delvecchio G. et al., Aust N Z J Psychiatry. 2018 Dec 13:4867418815976. doi: 10.1177/0004867418815976
- [Background] Neueder A. et al, J Mol Biol. 2018 Dec 29; S0022-2836(18)31287-7. doi: 10.1016/j.jmb.2018.12.012.
- [Background] Belzil VV, Gendron TF, Petrucelli L. RNA-mediated toxicity in neurodegenerative disease. Mol Cell Neurosci. 2013 Sep;56:406-19. doi: 10.1016/j.mcn.2012.12.006. Epub 2012 Dec 29. PMID 23280309
- [Background] Rademakers R, Eriksen JL, Baker M, Robinson T, Ahmed Z, Lincoln SJ, Finch N, Rutherford NJ, Crook RJ, Josephs KA, Boeve BF, Knopman DS, Petersen RC, Parisi JE, Caselli RJ, Wszolek ZK, Uitti RJ, Feldman H, Hutton ML, Mackenzie IR, Graff-Radford NR, Dickson DW. Common variation in the miR-659 binding-site of GRN is a major risk factor for TDP43-positive frontotemporal dementia. Hum Mol Genet. 2008 Dec 1;17(23):3631-42. doi: 10.1093/hmg/ddn257. Epub 2008 Aug 21. PMID 18723524
- [Background] Galimberti D, Villa C, Fenoglio C, Serpente M, Ghezzi L, Cioffi SM, Arighi A, Fumagalli G, Scarpini E. Circulating miRNAs as potential biomarkers in Alzheimer's disease. J Alzheimers Dis. 2014;42(4):1261-7. doi: 10.3233/JAD-140756. PMID 25024331
- [Background] Fenoglio C, Ridolfi E, Galimberti D, Scarpini E. An emerging role for long non-coding RNA dysregulation in neurological disorders. Int J Mol Sci. 2013 Oct 14;14(10):20427-42. doi: 10.3390/ijms141020427. PMID 24129177
- [Background] Ludwig B, Dwivedi Y. Dissecting bipolar disorder complexity through epigenomic approach. Mol Psychiatry. 2016 Nov;21(11):1490-1498. doi: 10.1038/mp.2016.123. Epub 2016 Aug 2. PMID 27480490
- [Background] Jin XF, Wu N, Wang L, Li J. Circulating microRNAs: a novel class of potential biomarkers for diagnosing and prognosing central nervous system diseases. Cell Mol Neurobiol. 2013 Jul;33(5):601-13. doi: 10.1007/s10571-013-9940-9. Epub 2013 Apr 30. PMID 23633081
- [Background] Fries GR, Walss-Bass C, Soares JC, Quevedo J. Non-genetic transgenerational transmission of bipolar disorder: targeting DNA methyltransferases. Mol Psychiatry. 2016 Dec;21(12):1653-1654. doi: 10.1038/mp.2016.172. Epub 2016 Oct 4. No abstract available. PMID 27698432
- [Background] Ghidoni R, Paterlini A, Albertini V, Glionna M, Monti E, Schiaffonati L, Benussi L, Levy E, Binetti G. Cystatin C is released in association with exosomes: a new tool of neuronal communication which is unbalanced in Alzheimer's disease. Neurobiol Aging. 2011 Aug;32(8):1435-42. doi: 10.1016/j.neurobiolaging.2009.08.013. Epub 2009 Sep 20. PMID 19773092
- [Background] Sanacora G, Treccani G, Popoli M. Towards a glutamate hypothesis of depression: an emerging frontier of neuropsychopharmacology for mood disorders. Neuropharmacology. 2012 Jan;62(1):63-77. doi: 10.1016/j.neuropharm.2011.07.036. Epub 2011 Aug 3. PMID 21827775
- [Background] Jun C, Choi Y, Lim SM, Bae S, Hong YS, Kim JE, Lyoo IK. Disturbance of the glutamatergic system in mood disorders. Exp Neurobiol. 2014 Mar;23(1):28-35. doi: 10.5607/en.2014.23.1.28. Epub 2014 Mar 27. PMID 24737937